CLINICAL TRIAL: NCT05666882
Title: HIV-IC: Effect on the HIV Diagnosis Rates of Integration of AIDS Defining and Indicator Conditions Into the Hospital Information Systems (HIS): 2 Phase, Multicenter Retrospective Study
Brief Title: Effect on the HIV Diagnosis Rates of Integration of AIDS Indicator Conditions Into the Hospital Information Systems
Acronym: HIV-IC
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Ankara University (Other)
Responsible Party: Principal Investigator, Ilker Kurkcu, Infectious Diseases Department, Ankara University
Other Study IDs: HIVIC
Record Dates: First submitted 2022-12-16; First posted 2022-12-28 (Actual); Last update posted 2022-12-28 (Actual); Status verified 2022-12

CONDITIONS: HIV Infections
MeSH Terms: conditions — HIV Infections

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: Non-interventional — Non-interventional

SUMMARY:
to describe the change in the number of HIV diagnosis before and after the integration of the indicator conditions and diseases to hospital automation system

DETAILED DESCRIPTION:
Scientific Basis/Rationale The HIV infection was first diagnosed in our country in 1985, and the number of the patients diagnosed with this infection has been gradually increasing since then. The number of these patients was found 21.520 in December 2018. Having CD4 cell count <350 cell/mm3 at the time of diagnosis or having an AIDS defining illness regardless of CD4 count has been defined as late diagnosis. 48-52% of HIV-positive cases have been shown to receive late diagnosis in the studies conducted in our country. It is being reported that there are no strategies of HIV screening for risky individuals and a significant part of the patients receive HIV diagnosis accidentally or during differential diagnosis of certain diseases. In the patients having late diagnosis, the treatment response is low and slow whereas progression to AIDS and death rates are high. The patients who could not be diagnosed also contribute to spread of the infection in the society. Therefore, it is significant that these patients should have early diagnosis and thus they could start treatment at the early phases of the infection in order to keep the disease under control. Hypothesis In the studies, it was reported that most of the patients with late diagnosis were the patients who were not defined to have a risk of HIV infection, although these patients had a number of applications to the healthcare centers before the diagnosis of the disease, HIV infection was not considered because they were not in the risky patient group and no tests were requested; therefore, the opportunities of the diagnosis could be missed. Diseases and the indicator conditions for which HIV test should be requested other than AIDS descriptive diseases are also identified in the studies conducted. The objectives of this study include studying the indicator conditions and diseases for which HIV test should be requested, determining the ratio of HIV test requests related to these conditions and diseases, integrating these diseases into the automation systems used in the hospitals and increasing the rate of HIV diagnosis by this means, prevention of missing diagnosis opportunities and raising awareness on this issue.

Primary Objective Change in the number of HIV diagnosis before and after the integration of the indicator conditions and diseases to hospital automation system Secondary Objectives Change in the number of HIV test requests before and after the integration of the indicator conditions and diseases to hospital automation system Assessment of CD4 levels at the time of diagnosis before and after the integration of the indicator conditions and diseases to hospital automation system Study Design and Research Methods This study has been designed as a multi-center retrospective cohort study. The indicator conditions and diseases for which HIV test should be requested will be recorded from the automation systems of the hospitals, and the rate of HIV test requests and rate of HIV positivity when the test was requested will be recorded for the all patients applied to hospital retrospectively for the past 6 months. For this period, due to retrospective design, physicians working at the hospitals do not have any information about the study. After the necessary approvals the indicator conditions and diseases for which HIV test should be requested shall be integrated into the hospitals automation systems and a warning stating that HIV test should be requested at the moment when these diseases and conditions are diagnosed shall pop-up. All the physicians working at the hospitals shall be notified of this activation by means of a letter. After this activation, 6 months later second retrospective step (phase) will start that, we will record the indicator conditions and diseases for which HIV test should be requested, and the rate of HIV test requests and the rate of HIV positivity when the test is requested will be recorded. During the study, the information obtained from the hospital automation system including age, gender, date of diagnoses, CD4 cell counts at the time of diagnoses, the HIV RNA levels, immigration status, concomitant diseases, and the residential area of all patients diagnosed with HIV infection shall be recorded on the appropriate forms. The characteristics of the patients that are diagnosed due to the indicator conditions and diseases for which HIV test should be requested shall be compared with the patients that are diagnosed due to other reasons. The HIV infection diagnoses rates during the two phases of the study shall also be compared. Furthermore, the patients shall be evaluated according to their CD4 counts at the time of the diagnosis, and shall be divided into two groups of patients as late diagnoses or not. We shall evaluate whether or not there is a difference regarding the rate of the patients with late diagnoses during the two phases of the study, and both groups shall be compared with respect to receiving late diagnosis factors.

The ethical approval of the study shall be obtained from the Ethical Committee of Ankara Training and Research Hospital. The centers participating in the study will obtain their approval to participate to the study from the centers where they work, using the ethical approval obtained form Ankara Training and Research Hospital. Each hospital will be responsible for the arrangements that must be made regarding the hospital automation system.

ELIGIBILITY:
Inclusion Criteria:

* All patients who apply to hospital to any clinic will be screened

Exclusion Criteria:

* Due to design of trial there will not be any exclusion criteria since all patients will be screened

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: All patients who apply to hospital to any clinic will be screened
Sampling Method: Non-Probability Sample
Enrollment: 10000 (Estimated)
Dates: Start 2022-06-01 (Actual); Primary Completion 2023-12-30 (Estimated); Study Completion 2024-02-28 (Estimated)

PRIMARY OUTCOMES:
Change in the number of HIV diagnosis before and after the integration of the indicator conditions and diseases to hospital automation system | Through study completion, an average of 18 months
  Change in the number of HIV diagnosis before and after the integration of the indicator conditions and diseases to hospital automation system

CONTACTS AND LOCATIONS:
Overall Officials: ilker kurkcu, Study Chair — Sentez-CRO
Locations (1):
- Ankara Eğitim ve Araştırma Hastanesi, Ankara, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No